CLINICAL TRIAL: NCT01239602
Title: The Variation of Movement Related Cortical Potential, Cortico-cortical Inhibition, and Motor Evoked Potential in Intracerebral Implantation of Antologous Peripheral Blood Stem Cells(CD34)in Old Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University Hospital
Other Study IDs: DMR99-IRB-200
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Stroke
Keywords: changes in cortical excitability in subjects with chronic stroke after stem cell therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Normal control
- with Stem cell therapy plus G-CSF
- G-CSF along

SUMMARY:
Stem cell theray in old stroke patients is a study to treat stroke patients approved before in our hospital. We recruit these patients who received stem cell therapy and completed the study. We adopted movement-related cortical potential,and cortico-cortical inhibition to assess the stroke patients with or without stem cell therapy. Further analyzing the correlation of the motor related cortical potential and cortico-cortical inhibition among them. We wanted to find out if there are changes in cortical excitability in subjects with chronic stroke after stem cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.old cerebral infarction (middle cerebral artery territory as documented on the T2 weight image [T2WI] of MRI) 2.between 6 months and 5 years of onset 3.National Institute of Health stroke scale (NIHSS) of between 9 and 20.

Exclusion Criteria:

* 1.Seizure history 2. Pacemaker insertion

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 36 patients suffered from old cerebral infarction (middle cerebral artery territory as documented on the T2 weight image [T2WI] of MRI) between 6 months and 5 years of onset who had initial scores on the National Institute of Health stroke scale (NIHSS) of between 9 and 20.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan